CLINICAL TRIAL: NCT00658463
Title: Effects of Rosuvastatin on the, in Vivo, Kinetic of VLDL apoB, IDL apoB, LDL apoB and HDL apoA1, Using Stable Isotopes, in Type 2 Diabetic Patients
Brief Title: Effects of Rosuvastatin on the, in Vivo, Kinetic of apoB and apoA1, Using Stable Isotopes, in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Prof. Bruno Vergès, Centre Hospitalier Universitaire Dijon
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFSSAPS 041348
Record Dates: First submitted 2008-04-02; First posted 2008-04-15 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes
Keywords: Diabetes; Triglycerides; HDL-cholesterol; kinetic; rosuvastatin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The study is designed with a one-month steady state period with placebo then on a cross-over design with two 6-week periods of placebo or rosuvastatin (20 mg). An in vivo kinetic study will be performed at the end of each 6-week period.
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator): The study is designed with a one-month steady state period with placebo then on a cross-over design with two 6-week periods of placebo or rosuvastatin (20 mg). An in vivo kinetic study will be performed at the end of each 6-week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — rosuvastatin 20 mg/day during 6 weeks versus placebo during 6 weeks in a cross-over design
  Other Names: CRESTOR (brand name for rosuvastatin)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Statins have been shown to reduce significantly the risk for cardiovascular events in patients with type 2 diabetes and statin therapy is largely recommended in this high cardiovascular risk population. However, a residual cardiovascular risk is observed in patients with type 2 diabetes treated by statins. This may be due to the fact that statins do not correct all lipid abnormalities associated with diabetic dyslipidaemia, such as hyperTG and low HDL-cholesterol.

Rosuvastatin is a statin which, in addition to its efficacy to reduce LDL-cholesterol, has been show to decrease significantly plasma triglycerides. However, the effects of rosuvastatin on triglyceride rich lipoproteins and HDL remains unknown. The purpose of this study is to analyze the effect rosuvastatin 20 mg on the metabolism of triglyceride rich lipoproteins and HDL in patients with Type 2 diabetes using and in vivo kinetic study of VLDL1-apoB,VLDL2-apoB,IDL-apoB and HDL-apoA1.

DETAILED DESCRIPTION:
This is a randomized, double blinded, placebo-controlled, monocentric, cross-over study with two 6-week periods of placebo or rosuvastatin. Subjects will enter a one month placebo lead-in period after which they will be eligible for rosuvastatin 20 mg or placebo for two 6-week periods.

An in vivo kinetic study will be performed with stable isotopes (13C leucine) in type 2 diabetic patients (n=8) before and after a 6-week period of rosuvastatin (20mg) therapy. The study is design with a one-month steady state period with placebo then on a cross-over design with two 6-week periods of placebo or rosuvastatin (20 mg. An in vivo kinetic study will be performed at the end of each 6-week period.

The kinetic studies performed, in each patient, will assess the production rates and fractional rates of VLDL1-apoB, VLDL2-apoB, IDL-apoB, LDL-apoB and HDL-apoA-I.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Type 2 diabetic patients (age: 30 to 75 years) treated by one or two oral agents at fixed dose (sulfonylureas, metformin, alpha glucosidase inhibitors) for at least 6 months
* Fasting triglycerides >= 150 mg/dl
* HDL-C < 40 mg/dl in men and < 50 mg/dl in women (NCEP ATPIII lipid criteria for the metabolic syndrome)
* Patients not receiving hypolipidemic agents since at least 6 months
* Diabetic patients with stable HbA1c during the last 6 months
* Subjects willing to follow all study procedures including attendance at clinic for scheduled study visits and compliance with study treatment regimen

Exclusion Criteria:

* HbA1c > 9 %
* LDL-C > 190 mg/dl
* Known heterozygous or homozygous familial hypercholesterolaemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia
* Documented secondary hypercholesterolaemia of any cause
* History of serious adverse effect or hypersensitivity reactions to other HMG-CoA reductase inhibitors, in particular any history of myopathy
* Pregnant women, women who are breast feeding and women of childbearing potential who are not using chemical or mechanical contraception (prescription oral contraceptives, abstinence, condoms with spermicide, surgical sterilisation, diaphragm with spermicide or intrauterine device) or have positive pregnancy test
* History of malignancy, except subjects who have been disease free for more than 10 years or whose only malignancy has been basal or squamous cell skin carcinoma. Women with a history of cervical dysplasia should be excluded unless 3 consecutive normal cervical smears have subsequently been recorded before entry into the study
* History of alcohol and/or drug abuse
* Active liver disease or hepatic dysfunction as defined by elevations of AST or ALT * 2 times the ULN. In this case, a second determination of hepatic tests will be performed after one week. If the dysfunction is confirmed, the subject must not be included in the study
* Patient with acromegaly or Cushing syndrome
* Patient receiving insulin treatment
* Use of drugs known to affect lipid metabolism: corticoids, retinoids, antiproteases, estrogens, cyclosporin, glitazones, statins other than rosuvastatin, fibrates, cholestyramine, nicotinic acid, omega 3 or phytosterols
* Renal impairment as defined by creatinine clearance < 30 ml/min.
* Unstable angina or manifestation of severe atherosclerosis.
* Uncontrolled hypertension defined as either resting diastolic blood pressure of >95mmHg or resting systolic blood pressure of >200 mmHg.
* Unexplained serum CK > 3 times ULN (eg. not due to recent trauma, intramuscular injections, heavy exercise, etc).
* Participation in another investigational drug trial within 4 weeks prior to randomization.
* Subjects with serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the trial.
* Subjects with serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Fractional Catabolic Rates (FCR)of VLDL1-apoB, VLDL2-apoB, IDL-apoB, LDL-apoB and HDL-apoA-I | At the end of each treatment period (rosuvastatin or placebo)

SECONDARY OUTCOMES:
Production Rates (PR) of VLDL1-apoB, VLDL2-apoB, IDL-apoB, LDL-apoB and HDL-apoA-I | At the end of each treatment period (rosuvastatin or placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vergès, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- Centre Hospitalier Universitaire de Dijon, Dijon, France

REFERENCES:
- [Derived] Verges B, Florentin E, Baillot-Rudoni S, Monier S, Petit JM, Rageot D, Gambert P, Duvillard L. Effects of 20 mg rosuvastatin on VLDL1-, VLDL2-, IDL- and LDL-ApoB kinetics in type 2 diabetes. Diabetologia. 2008 Aug;51(8):1382-90. doi: 10.1007/s00125-008-1046-4. Epub 2008 Jun 5. PMID 18535816